CLINICAL TRIAL: NCT04852003
Title: A Phase Ⅲ, Randomized, Double-blind, Placebo- and Active-controlled Study of SHR0410 Injection for the Treatment of Pain After Endoscopic Surgery of the Lower Abdominal
Brief Title: A Trial of SHR0410 Injection for the Treatment of Pain After Endoscopic Surgery of the Lower Abdominal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0410-301
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: SHR0410 injection compared with placebo and morphine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR0410 Injection (Experimental)
  Interventions: Drug: SHR0410 Injection
- Placebo for SHR0410 Injection (Placebo Comparator)
  Interventions: Drug: Placebo
- Morphine (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: SHR0410 Injection — SHR0410 Injection
  Arms: SHR0410 Injection
Drug: Placebo — Placebo for SHR0410 Injection
  Arms: Placebo for SHR0410 Injection
Drug: Morphine — Morphine
  Arms: Morphine

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR0410 injection for the treatment of pain after endoscopic surgery of the lower abdominal.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia endoscopic surgery of the lower abdominal
3. Male or female
4. Meet the body mass index standard
5. Conform to the ASA Physical Status Classification

Exclusion Criteria

1. Subjects with a history of difficult airway
2. Subjects with a history of mental illness
3. Subjects with a history of cognitive impairment epilepsy
4. Subjects with a history of myocardial infarction or unstable angina pectoris
5. Subjects with atrioventricular block or cardiac insufficiency
6. Subjects with a history of ischemic stroke or transient ischemic attack
7. Subjects with poor blood pressure control after medication
8. Subject with a history of substance abuse and drug abuse
9. Abnormal values in liver function
10. Subjects with an oxygen saturation below 90% on room air
11. Allergic to drugs that may be used during the study
12. Pregnant or nursing women
13. No birth control during the specified period of time
14. Participated in clinical trials of other drugs (received experimental drugs)
15. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
The area under the curve of pain intensity over 24 hours | 24-hours
  Pain intensity will be evaluated using an 11-point (0-10) numeric rating scale (NRS), with higher numbers indicating a higher pain intensity, administered over 24 hours.

SECONDARY OUTCOMES:
Total consumption of remedial analgesics from 0h to 24h | 24-hours
  Total consumption of IV morphine
Participant ' satisfaction score for analgesia treatment | 24-hours
  Participants recalled the postoperative analgesia effect and rated their satisfaction on a scale of 0 to 10, with 0 representing dissatisfied and 10 representing very satisfied.
Investigator satisfaction score for analgesia treatment | 24-hours
  Postoperative analgesia was evaluated by investigators. The scale ranges from 0 to 10, with 0 being dissatisfied and 10 being very satisfied.
Frequency and severity of adverse events | Day 4（or early termination on Day 3）
  Assessed by monitoring of adverse events. Participants with adverse events found to be related to the study drug will be compared to those receiving placebo or active comparator.
Safety as assessed by vital signs | Day 4（or early termination on Day 3）
  Changes in vital signs such as body temperature, blood pressure, heart rate will be assessed at specified times.
Safety as assessed by laboratory evaluations | Day 4（or early termination on Day 3）
  Assessed by laboratory evaluations at specified times. Participants with clinically significant lab values will be compared to those receiving placebo or active comparator.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China